CLINICAL TRIAL: NCT02458651
Title: An Observational Study of Patients With Newly Diagnosed Unresectable Stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC) in China
Brief Title: Disease Characteristics, Treatment Patterns and Clinical Outcomes in Patients With Newly Diagnosed Unresectable Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) in China
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: YO29443
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Non-Small Cell Lung Cancer, Lung Cancer, Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Tier 1 and North: Site as described by tier level of the city where the site is located and by geographical location: Tier 1 city in northern region of China
  Interventions: Other: No intervention
- Tier 1 and South: Site as described by tier level of the city where the site is located and by geographical location: Tier 1 city in southern region of China
  Interventions: Other: No intervention
- Tier 2 and Middle: Site as described by tier level of the city where the site is located and by geographical location: Tier city in middle region of China
  Interventions: Other: No intervention
- Tier 2 and North: Site as described by tier level of the city where the site is located and by geographical location: Tier 2 city in northern region of China
  Interventions: Other: No intervention
- Tier 2 and South Eastern: Site as described by tier level of the city where the site is located and by geographical location: Tier 2 city in south eastern region of China
  Interventions: Other: No intervention
- Tier 2 and South Western: Site as described by tier level of the city where the site is located and by geographical location: Tier 2 city in south western region of China
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
The purpose of this observational study is to describe patient and disease characteristics as well as treatment patterns in Chinese patients with unresectable stage IIIB or IV non-small cell lung cancer (NSCLC). In addition, this study characterizes the clinical outcomes for various populations of patients defined by clinical and tumor characteristics, treatment patterns, and hospital category defined by city tier and geographic region.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, unresectable Stage IIIB or IV non-small cell lung cancer (NSCLC)
* Received at least one anti-cancer treatment targeting unresectable Stage IIIB or IV NSCLC in the study site after study initiation
* Radiographic evidence of disease

Exclusion Criteria:

* Prior systematic treatment for unresectable Stage IIIB or IV non-small cell lung cancer (NSCLC)
* Participation in any anti-cancer, regimen-specified clinical study of first-line treatment for unresectable Stage IIIB or IV NSCLC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with newly diagnosed, unresectable Stage IIIB or IV non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 1378 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Demographic and Socio-Behavioral Characteristics | At enrollment
Medical History Characteristics | At enrollment
Score Tumor Characteristics Based on Tumor Histology, Stage, Grade, and Lung Cancer Molecular Profile | At enrollment, during quarterly and semi-annual follow up and at end of study up to 1.5 years
Grade of Eastern Cooperative Oncology Group (ECOG) Performance Status | At enrollment, during quarterly and semi-annual follow up and at end of study up to 1.5 years
Treatment Patterns of First-Line and Subsequent Treatments | At enrollment, during quarterly and semi-annual follow up and at end of study up to 1.5 years
Progression-Free Survival (PFS) | From enrollment to end of study up to 1.5 years
Overall Survival (OS) | From enrollment to end of study up to 1.5 years

SECONDARY OUTCOMES:
Score Health Economic Status Based on Household Income, Diagnosis and Treatment Costs, and Insurance Coverage | At enrollment, during quarterly and semi-annual follow up and at end of study up to 1.5 years
Percentage of Serious Adverse Events (SAEs) | From enrollment to end of study up to 1.5 years
Percentage of Adverse Events (AEs) | From enrollment to end of study up to 1.5 years
Percentage of Non-Serious AEs of Special Interest (AESIs) | From enrollment to end of study up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- China (11):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - the First Hospital of Jilin University, Changchun
  - Sichuan Provincial Cancer Hospital, Chengdu
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an